CLINICAL TRIAL: NCT03831204
Title: Systolic Time Intervals a Pronostic Tool of Heart Failure in Emergency Departement
Brief Title: Systolic Time Intervals a Prognostic Tool of Heart Failure in Emergency Departement (STI/AHF)
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Other Study IDs: STI in AHF prognostic
Record Dates: First submitted 2018-07-06; First posted 2019-02-05 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Dyspnea; Heart Failure
Keywords: impedance; dyspnea; AHF; BNP; EFFECT; GWTG-HF
MeSH Terms: conditions — Dyspnea; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AHF/HFpEF: AHF with preserved ejection fraction Acoustic cardiography was performed for all participants using the BIOPAC Prognostic scores were calculated for every patient
  Interventions: Device: biopac; Diagnostic Test: prognostic scores
- AHF/HFrEF: AHF with reduced ejection fraction Acoustic cardiography was performed for all participants using the BIOPAC Prognostic scores were calculated for every patient
  Interventions: Device: biopac; Diagnostic Test: prognostic scores

INTERVENTIONS:
Device: biopac — Acoustic cardiography was performed for all participants using the BIOPAC system with "Student Lab" software version 3.7.2. An electrocardiogram was obtained by two electrodes placed at the right upper limb and the lower left limb. Simultaneously heart sounds were recorded with a specific sensor placed at the mitral focus.
Diagnostic Test: prognostic scores — Effect and GWTGHF were calculated for every patient

SUMMARY:
The performance of STIs and clinical scores alone and their combination to predict short term prognosis of acute decompensated heart failure.

DETAILED DESCRIPTION:
Acute heart failure is a leading cause of hospitalization and death.Prediction of these adverse events is still challenging.

STI is an old technique based on the recording of two parameters: electrocardiogram and phonocardiogram, and from them measuring the different systolic intervals:

pre-ejection period (PEP),electro-mechanic activation time (EMAT), Left ventricular ejection time (LVET) and systolic time ratio (RTS) were measured.

The aim of these study is to demonstrate whether systolic time intervals (STIs) can improve clinical scores EFFECT (Enhanced Feedback for Effective Cardiac Treatment) and GWTG-HF (Get With the Guidelines-Heart Failure) for predicting 30 day mortality and readmission in patients with acute decompensated heart failure (ADHF) in the ED.

ELIGIBILITY:
Inclusion Criteria:

* non traumatic dyspnea
* age more than 18 years old.

Exclusion Criteria:

* ECG diagnostic for acute myocardial infarction
* ischemic chest pain within the prior 24 hours
* history of a heart transplant
* pericardial effusion
* chest wall deformity suspected of causing dyspnea
* coma
* shock,Mechanical Ventilation, vasopressor drugs
* arrhythmia serious and sustained,
* pace maker
* severe mitral valve disease,
* severe pulmonary arterial hypertension
* renal failure with creatinine >350micromol/l

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all patients aged more than 18 years admitted to the ED with the diagnosis of acute decompensated heart failure
Sampling Method: Non-Probability Sample
Enrollment: 642 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
compare the STIs prognostic performance against clinical scores | 30 days
  the area under ROC curve of the Systolic Time Intervals compared to the one of the EFFECT and GWTG HF scores

SECONDARY OUTCOMES:
compare the STI prognostic performance between HFpEF and HFrEF patients | 30 days
  compare the STI prognostic performance between HFpEF and HFrEF patients using the area under curve estimation of the ROC curve of the three systolic time intervals (PEP;EMAT measured in milliseconds,and PEP/EMAT) of the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Pr, Principal Investigator — University hospital of Monastir
Locations (1):
- Emergency department of university hospital Fattouma Bourguiba of Monastir Monastir, Monastir Tunisia, Monastir, Tunisia

REFERENCES:
- See also: official department website — http://www.urgencemonastir.com